CLINICAL TRIAL: NCT05375760
Title: A Phase II Randomized, Open-label, Multicenter, Dose-ranging Study in Adults and Pediatric Individuals ≥ 12 Years of Age to Assess the Safety, Immunogenicity, Pharmacokinetics, and Pharmacodynamics of AZD7442, a Combination Product of Two Monoclonal Antibodies (Tixagevimab and Cilgavimab), for Pre-exposure Prophylaxis of COVID-19
Brief Title: A Randomized, Open-label, Dose-ranging Study in Adults and Pediatric Individuals ≥ 12 Years of Age to Assess the Safety, Immunogenicity, Pharmacokinetics, and Pharmacodynamics of AZD7442, for Pre-exposure Prophylaxis of COVID-19
Acronym: ENDURE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor terminated after review of FDA's request to halt further dosing (30Mar2023) given that AZD7442 is not active against >99% of the currently circulating SARS-CoV-2 variants in the USA, the benefit risk assessment may not be favorable
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: D8850C00010; 2022-001014-20 (EudraCT Number)
Record Dates: First submitted 2022-05-16; First posted 2022-05-17 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-09

CONDITIONS: Coronavirus Disease 2019 (COVID-19)
Keywords: ENDURE
MeSH Terms: conditions — COVID-19 | interventions — cilgavimab and tixagevimab drug combination; tixagevimab; cilgavimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Other): 600 mg AZD7442 following 300 mg AZD7442 every 3 months (5 doses totally)
  Interventions: Biological: AZD7442 (tixagevimab [AZD8895] + cilgavimab [AZD1061])
- Arm B (Other): 1200mg AZD7442 following 600 mg AZD7442 every 6 months (3 doses totally)
  Interventions: Biological: AZD7442 (tixagevimab [AZD8895] + cilgavimab [AZD1061])

INTERVENTIONS:
Biological: AZD7442 (tixagevimab [AZD8895] + cilgavimab [AZD1061]) — Arm A - Day 1:
  600 mg AZD7442 administered sequentially as a 3 mL IM injection containing 300 mg tixagevimab (AZD8895) and a 3 mL IM injection containing 300 mg cilgavimab (AZD1061), one injection in each gluteal region.
  Arm A - Days 92, 183, 274, 365:
  300 mg AZD7442 administered sequentially as a 1.5 mL IM injection containing 150 mg tixagevimab (AZD8895) and a 1.5 mL IM injection containing 150 mg cilgavimab (AZD1061), one injection in each gluteal region.
  Arms: Arm A
Biological: AZD7442 (tixagevimab [AZD8895] + cilgavimab [AZD1061]) — Arm B - Day 1:
  1200 mg AZD7442 (600 mg tixagevimab [AZD8895] and 600 mg cilgavimab [AZD1061]) administered by IV infusion.
  Arm B - Days 183, 365:
  600 mg AZD7442 administered sequentially as a 3 mL IM injection containing 300 mg tixagevimab (AZD8895) and a 3 mL IM injection containing 300 mg cilgavimab (AZD1061), one injection in each gluteal region.
  Arms: Arm B

SUMMARY:
A Phase II Randomized, Open-label, Multicenter, Dose-ranging Study in Adults and Pediatric Individuals ≥ 12 years of Age to Assess the Safety, Immunogenicity, Pharmacokinetics, and Pharmacodynamics of AZD7442, a Combination Product of Two Monoclonal Antibodies (Tixagevimab and Cilgavimab), for Pre-exposure Prophylaxis of COVID-19

DETAILED DESCRIPTION:
AZD7442, a combination of 2 monoclonal antibodies (tixagevimab [investigational name, AZD8895] and cilgavimab [investigational name, AZD1061]), is being developed for the prophylaxis and treatment of coronavirus disease 2019 (COVID-19).

This Phase II dose-ranging study will investigate the safety, immunogenicity, pharmacokinetic (PK), and pharmacodynamic (PD) profiles of AZD7442 repeat dosing regimens for preexposure prophylaxis of COVID-19 in adults and pediatric individuals (≥ 12 years of age weighing at least 40 kg), who are moderately to severely immunocompromised.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent as described in Appendix A which includes compliance with the requirements and restrictions listed in the ICF and in this protocol. For pediatric participants: informed assent is to be provided by the participant; informed consent must be provided by the participant's legal guardian 2. Ensure that participants who are considered by the Investigator clinically unable to consent at screening and who are entered into the study by the consent of a legally acceptable representative show evidence of assent, as applicable in accordance with local regulations.

3. Participant must be an adult (≥ 18 years of age) or pediatric individual (≥ 12 to < 18 years of age weighing ≥ 40 kg) at the time of signing the ICF or assent (for pediatric participants).

4. Individuals with medical conditions or treatments that may result in moderate to severe immune compromise or an inadequate immune response to COVID-19 vaccination include but are not limited to:

1. Active treatment for solid tumor and hematologic malignancies.
2. Receipt of solid-organ transplant and taking immunosuppressive therapy.
3. Receipt of chimeric antigen receptor T-cell or hematopoietic stem cell transplant (within 2 years of transplantation or taking immunosuppression therapy).
4. Moderate or severe primary immunodeficiency (eg, DiGeorge syndrome, Wiskott-Aldrich syndrome).
5. Advanced or untreated HIV infection (people with HIV and history of CD4 cellcounts < 200/mm3, history of an AIDS-defining illness without immune reconstitution, or clinical manifestations of symptomatic HIV).
6. Active treatment with systemic high-dose corticosteroids (ie, ≥ 20 mg prednisone or equivalent per day when administered for ≥ 2 weeks), alkylating agents, antimetabolites, transplant-related immunosuppressive drugs, cancer chemotherapeutic agents classified as severely immunosuppressive, tumor necrosis factor blockers, and other biologic agents that are immunosuppressive or immunomodulatory (eg, B-cell depleting agents).

   5 Documented negative SARS-CoV-2 RT-PCR test from an NP specimen collected ≤ 3 days prior to Day 1 or a negative SARS-CoV-2 rapid antigen test from an NP specimen at screening.

   Exclusion Criteria:
   1. Any clinical signs and symptoms consistent with COVID-19, eg, fever, dry cough, dyspnea, sore throat, fatigue for ≥ 5 days or confirmed COVID-19 infection by appropriate laboratory test within 28 days prior to screening. Prior COVID-19 infection is not an exclusion.
   2. History or current hospitalization for worsening disease during the one month prior to screening, with no change in condition at the time of study enrollment as judged by the Investigator.
   3. Current need for hospitalization or immediate medical attention in a clinic or emergency room service in the clinical opinion of the Investigator.
   4. Previous hypersensitivity, infusion-related reaction, or severe adverse reaction following administration of a mAb.
   5. Known history of allergy to any component of the IMP formulation.
   6. History of clinically significant bleeding disorder (eg, factor deficiency, coagulopathy, or platelet disorder), or prior history of significant bleeding or bruising following IV infusions or venepuncture.
   7. Any other significant disease, disorder, or finding that may significantly increase the risk to the participant because of participation in the study, affect the ability of the participant to participate in the study, or impair interpretation of the study data
   8. Any co-morbidity requiring surgery within 7 days prior to study entry, or that is considered life-threatening in the opinion of the Investigator within 30 days prior to study entry.

   9 Any prior receipt of investigational or licensed mAb or other biologic indicated for the prevention or treatment of SARS-CoV-2 or COVID-19 within 5 half-lives prior to screening or expected administration immediately after enrollment.

   10 Have received a COVID-19 vaccination ≤ 14 days before Day 1 or plan to receive a COVID-19 vaccination ≤ 14 days after Day 1 (Such participants can subsequently be included in the study once they have reached > 14 days after their last dose of vaccine).

   11 Receipt of convalescent COVID-19 plasma treatment within 90 days prior to screening.

   12 Receipt of any IMP in the preceding 90 days or 5 half-lives, whichever is longer, or expected receipt of IMP during the period of study follow-up, or concurrent participation in another interventional study.

   13 Judgment by the Investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions, and requirements.

   14 For women only - currently pregnant (confirmed with positive pregnancy test) or breastfeeding.

   15 Previous randomization in the present study. 16 Blood drawn in excess of a total of 450 mL (1 unit) for any reason within 30 days prior to randomization.

   17 Employees of the Sponsor involved in planning executing, supervising, or reviewing the AZD7442 program, clinical study site staff, or any other individuals involved with the conduct of the study, or immediate family members of such individuals.

   18 In nations, states, or other jurisdictions that for legal or ethical reasons bar the enrollment of participants who lack capacity to provide their own informed consent, such subjects are excluded.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2023-10-04 (Actual); Study Completion 2023-10-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Research Site, Birmingham, Alabama
  - Research Site, Modesto, California
  - Research Site, Westminster, California
  - Research Site, Hollywood, Florida
  - Research Site, Lake City, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Ormond Beach, Florida
  - Research Site, Wesley Chapel, Florida
  - Research Site, West Palm Beach, Florida
  - Research Site, Chicago, Illinois
  - Research Site, St Louis, Missouri
  - Research Site, Knoxville, Tennessee
  - Research Site, Austin, Texas
  - Research Site, El Paso, Texas
  - Research Site, Annandale, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00010&attachmentIdentifier=6b2c1724-502c-49b0-96c6-f4b8875fa267&fileName=D8850C00010-SAP-_redacted.pdf&versionIdentifier=
- See also: redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00010&attachmentIdentifier=48cfe85b-3834-4ee2-b519-009d7d2eca78&fileName=D8850C00010-CSP_redacted.pdf&versionIdentifier=
- See also: redacted CRS Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D8850C00010&attachmentIdentifier=6070265d-3c05-4452-b3ef-f12f90ba58f3&fileName=D8850C00010-CSR-Synopsis_Redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The participants were screened and randomized from the USA. First subject in was on 09Jun2022 and the last subject last visit was 04Oct2023. Sponsor terminated the study after review of FDA's request to halt further dosing (30Mar2023) and subjects were terminated prior to 1 year dose given that AZD7442 is not active against >99% of the currently circulating SARS-CoV-2 variants in the USA, the benefit risk assessment may not be favorable.
Groups:
- AZD7442: 600 mg ONCE / 300mg Q3M: AZD7442 600 mg intramuscularly (IM) on Day 1 followed by 300 mg IM every 3 months (Q3M) for 12 months.
- AZD7442: 1200mg ONCE / 600mg Q6M: AZD7442 1200 mg intravenously (IV) on Day 1 followed by 600 mg IM every 6 months (Q6M) for 12 months.
Period: Overall Study
Arm/Group | AZD7442: 600 mg ONCE / 300mg Q3M | AZD7442: 1200mg ONCE / 600mg Q6M
Started | 125 | 126
Treated | 124 | 124
Completed | 0 | 0
Not Completed | 125 | 126
Not completed — Adverse Event | 1 | 0
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 6 | 6
Not completed — Withdrawal by Subject | 17 | 19
Not completed — Dosing halted by FDA | 96 | 100
Not completed — Not compliant with study visit | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Signed ICF addendum, however refused procedures | 1 | 0
Not completed — Participant moved | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set: participants who received IMP and classified according to the treatment they actually received.
Groups:
- AZD7442: 600mg ONCE / 300mg Q3M: AZD7442 600 mg intramuscularly (IM) on Day 1 followed by 300 mg IM every 3 months (Q3M) for 12 months.
- AZD7442: 1200 mg ONCE / 600mg Q6M: AZD7442 1200 mg intravenously (IV) on Day 1 followed by 600 mg IM every 6 months (Q6M) for 12 months.
- Total: Total of all reporting groups
Arm/Group | AZD7442: 600mg ONCE / 300mg Q3M | AZD7442: 1200 mg ONCE / 600mg Q6M | Total
Number analyzed (Participants) | 124 | 124 | 248
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (13.97) | 54.2 (14.85) | 55.7 (14.47)
Age, Customized [Number; unit: Participants]
  >=12 - <18 | 0 | 0 | 0
  >=18 - <65 | 86 | 98 | 184
  >=65 - <75 | 26 | 12 | 38
  >=75 - <80 | 9 | 7 | 16
  >=80 | 3 | 7 | 10
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Safety Analysis Set
  Participants
    Female | 65 | 67 | 132
    Male | 59 | 57 | 116
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Safety Analysis Set
  Participants
    Hispanic or Latino | 63 | 60 | 123
    Not Hispanic or Latino | 60 | 64 | 124
    Not reported | 1 | 0 | 1
    Unknown | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Population: Safety Analysis Set
  Participants
    White | 96 | 94 | 190
    Black or African American | 20 | 23 | 43
    Asian | 3 | 3 | 6
    American Indian or Alaska Native | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Multiple | 2 | 0 | 2
    Unknown | 1 | 0 | 1
    Not reported | 1 | 3 | 4
Screening result from Nasopharyngeal swab for SARS-CoV-2 RT-PCR [Count of Participants; unit: Participants]
  Negative | 124 | 124 | 248
  Positive | 0 | 0 | 0
Previous COVID-19 vaccination [Count of Participants; unit: Participants] — Administered prior to first IMP dose Population: The numbers in the different subcategories (row) are cumulative. So they do not sum up to the made categories
  Participants
    Yes | 26 | 19 | 45
    No | 98 | 105 | 203
Time since previous COVID-19 vaccination [Median (Inter-Quartile Range); unit: Days] — Partial COVID-19 vaccination dates with missing days were imputed at the last day of the month Population: Number of participants with a previous COVID-19 infection
  Days
    number analyzed (Participants) | 26 | 19 | 45
    (all) | 107.0 [79.0 to 305.0] | 205.0 [105.0 to 354.0] | 138.0 [85.0 to 320.0]
Smoking history [Count of Participants; unit: Participants]
  Current | 23 | 13 | 36
  Former | 28 | 24 | 52
  Never | 73 | 87 | 160
Number of pack years (Current or Former) [Mean (Standard Deviation); unit: percentages] — Population: Number of participants having current or former smoking history
  percentages
    number analyzed (Participants) | 51 | 37 | 88
    (all) | 18.9 (19.27) | 20.0 (18.74) | 19.3 (18.95)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 81.17 (20.764) | 83.27 (19.258) | 82.22 (20.013)
Height (cm) [Mean (Standard Deviation); unit: cm] | 168.18 (10.406) | 167.68 (9.946) | 167.93 (10.162)
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 28.66 (6.884) | 29.66 (6.582) | 29.16 (6.740)
Body Mass Index (kg/m^2) Category [Count of Participants; unit: Participants]
  < 25 | 32 | 26 | 58
  25 - <30 | 52 | 47 | 99
  30 - <35 | 25 | 29 | 54
  >= 35 | 15 | 22 | 37

OUTCOME MEASURES:

1. Primary Outcome: AEs, SAEs, and AESIs
Description: To evaluate the safety and tolerability of AZD7442
Time Frame: Safety data were recorded from the time of the first IMP administration throughout the study for an average safety follow up time of 48.85 weeks. This was shorter than the planned one of 105 weeks due to FDA's request to halt dosing.
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7442: 600mg ONCE / 300mg Q3M | AZD7442: 1200 mg ONCE / 600mg Q6M
Number analyzed (Participants) | 124 | 124
Participants
  Adverse Events | 84 | 66
  Serious Adverse Events | 13 | 10
  Adverse Events of Special Interest | 9 | 7

2. Primary Outcome: ADA in Serum Responses
Description: To evaluate the immunogenicity of AZD7442
Time Frame: Serum ADA were assessed through the treatment period at the specific timepoints: baseline, 29, 92, 121 (300mg Q3M arm only), 183, 212, 274, 365, 456 days or early discontinuation visit after the first IMP administration.
Population: ADA Evaluable Analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | AZD7442: 600mg ONCE / 300mg Q3M | AZD7442: 1200 mg ONCE / 600mg Q6M
Number analyzed (Participants) | 106 | 111
Participants | 1 | 3

3. Secondary Outcome: Serum AZD7442 Concentrations
Description: To evaluate the PK of AZD7442 in serum
Time Frame: Serum PK was assessed through the treatment period at the specific timepoints: day 1 post-dose (600mg Q6M arm only), 3, 11, 29, 92, 121 (300mg Q3M arm only), 183, 212, 274, 365 days or early discontinuation visit after the first IMP administration.
Population: PK Analysis Set
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | AZD7442: 600mg ONCE / 300mg Q3M | AZD7442: 1200 mg ONCE / 600mg Q6M
Number analyzed (Participants) | 107 | 116
ug/mL
  Day 1, Post-dose: number analyzed (Participants) | 0 | 91
  Day 1, Post-dose |  | 285.8539 (176.0959)
  Day 3: number analyzed (Participants) | 28 | 33
  Day 3 | 30.0089 (83.7707) | 165.1457 (196.9756)
  Day 11: number analyzed (Participants) | 28 | 33
  Day 11 | 45.5626 (53.9503) | 123.2505 (160.5606)
  Day 29: number analyzed (Participants) | 98 | 97
  Day 29 | 40.0381 (48.7457) | 105.8292 (76.5535)
  Day 92: number analyzed (Participants) | 98 | 106
  Day 92 | 27.9754 (48.9241) | 63.0711 (76.0487)
  Day 121: number analyzed (Participants) | 89 | 0
  Day 121 | 42.1820 (53.2624) |
  Day 183: number analyzed (Participants) | 97 | 102
  Day 183 | 23.8985 (58.4175) | 26.4300 (85.1380)
  Day 212: number analyzed (Participants) | 92 | 101
  Day 212 | 36.5360 (54.5622) | 60.5211 (44.6566)
  Day 274: number analyzed (Participants) | 89 | 96
  Day 274 | 24.3601 (59.3582) | 38.1694 (55.8293)
  Day 365: number analyzed (Participants) | 3 | 97
  Day 365 | 21.2009 (46.2521) | 17.2078 (91.1273)
  Confirmed Illness 1 Day 1: number analyzed (Participants) | 5 | 6
  Confirmed Illness 1 Day 1 | 36.2743 (30.3957) | 103.0573 (43.1944)
  Confirmed Illness 1 Day 14: number analyzed (Participants) | 6 | 7
  Confirmed Illness 1 Day 14 | 37.2795 (25.1834) | 79.1638 (29.7188)

4. Secondary Outcome: Changes From Baseline in GMTs Values in SARSCoV- 2 nAbs (Wild-type Assay)
Description: To determine anti severe acute respiratory coronavirus-2 neutralizing antibodies (anti-SARS-CoV 2 nAb) levels in serum after administration of AZD7442
Time Frame: SARSCoV-2 nAbs (Wild Type Assay) were assessed through the treatment period at these specific timepoints: baseline, 29, 92, 121 (300mg Q3M arm only), 183, 212, 274, 365 days or early termination visit after the first IMP administration.
Population: nAb Evaluable Analysis Set - Authentic Virus
Measure: Geometric Mean (Standard Deviation); unit: Titer
Arm/Group | AZD7442: 600mg ONCE / 300mg Q3M | AZD7442: 1200 mg ONCE / 600mg Q6M
Number analyzed (Participants) | 112 | 119
Titer
  Baseline Titer: number analyzed (Participants) | 112 | 111
  Baseline Titer | 203.5 (6.43) | 198.9 (7.70)
  Day 29 Titer: number analyzed (Participants) | 109 | 109
  Day 29 Titer | 1442.8 (1.88) | 3497.1 (2.10)
  Day 92 Titer: number analyzed (Participants) | 91 | 105
  Day 92 Titer | 1052.5 (2.22) | 2268.6 (2.30)
  Day 121 Titer: number analyzed (Participants) | 84 | 0
  Day 121 Titer | 1520.2 (1.97) |
  Day 183 Titer: number analyzed (Participants) | 84 | 96
  Day 183 Titer | 1209.8 (1.95) | 1337.9 (2.10)
  Day 212 Titer: number analyzed (Participants) | 81 | 90
  Day 212 Titer | 941.2 (2.08) | 1436.1 (1.78)
  Day 274 Titer: number analyzed (Participants) | 74 | 88
  Day 274 Titer | 488.5 (2.38) | 864.7 (1.98)
  Day 365 Titer: number analyzed (Participants) | 2 | 83
  Day 365 Titer | 482.1 (1.21) | 578.9 (2.21)

5. Secondary Outcome: Changes From Baseline in GMTs in SARSCoV- 2 nAbs (Pseudo Neutralization Assay)
Description: as for outcome 4
Time Frame: SARSCoV-2 nAbs (Pseudo Neutralization Assay) were assessed through the study at these specific timepoints: baseline, 29, 92, 121 (300mg Q3M arm only), 183, 212, 274, 365 days or early termination visit after the first IMP administration.
Population: nAb Evaluable Analysis Set - Pseudo Virus
Measure: Geometric Mean (Standard Deviation); unit: Titer
Arm/Group | AZD7442: 600mg ONCE / 300mg Q3M | AZD7442: 1200 mg ONCE / 600mg Q6M
Number analyzed (Participants) | 112 | 119
Titer
  Baseline Titer: number analyzed (Participants) | 94 | 97
  Baseline Titer | 1613.3 (7.96) | 1735.8 (8.35)
  Day 29 Titer: number analyzed (Participants) | 106 | 115
  Day 29 Titer | 32170.5 (1.86) | 111726.8 (1.75)
  Day 92 Titer: number analyzed (Participants) | 83 | 104
  Day 92 Titer | 13940.9 (1.88) | 38048.0 (1.73)
  Day 121 Titer: number analyzed (Participants) | 82 | 0
  Day 121 Titer | 23177.5 (1.87) |
  Day 183 Titer: number analyzed (Participants) | 79 | 93
  Day 183 Titer | 12018.5 (1.75) | 15554.6 (1.80)
  Day 212 Titer: number analyzed (Participants) | 77 | 94
  Day 212 Titer | 19353.3 (1.72) | 36519.3 (1.67)
  Day 274 Titer: number analyzed (Participants) | 69 | 79
  Day 274 Titer | 12816.8 (1.93) | 23583.5 (1.91)
  Day 365 Titer: number analyzed (Participants) | 2 | 76
  Day 365 Titer | 5068.4 (1.55) | 7155.4 (2.01)

6. Secondary Outcome: Changes From Baseline in GMFRs Values in SARSCoV- 2 nAbs (Wild-type Assay)
Description: as for outcome 4
Time Frame: as for outcome 4
Population: nAb Evaluable Analysis Set - Authentic Virus
Measure: Geometric Mean (Standard Deviation); unit: Fold rise
Arm/Group | AZD7442: 600mg ONCE / 300mg Q3M | AZD7442: 1200 mg ONCE / 600mg Q6M
Number analyzed (Participants) | 112 | 119
Fold rise
  Day 29 fold rise: number analyzed (Participants) | 105 | 106
  Day 29 fold rise | 6.87 (4.765) | 16.79 (6.429)
  Day 92 fold rise: number analyzed (Participants) | 87 | 101
  Day 92 fold rise | 4.32 (4.329) | 10.53 (6.362)
  Day 121 fold rise: number analyzed (Participants) | 83 | 0
  Day 121 fold rise | 6.53 (4.928) |
  Day 183 fold rise: number analyzed (Participants) | 80 | 93
  Day 183 fold rise | 5.29 (4.744) | 5.43 (5.122)
  Day 212 fold rise: number analyzed (Participants) | 77 | 88
  Day 212 fold rise | 4.09 (5.554) | 5.28 (6.243)
  Day 274 fold rise: number analyzed (Participants) | 71 | 83
  Day 274 fold rise | 1.96 (4.385) | 3.08 (5.820)
  Day 365 fold rise: number analyzed (Participants) | 2 | 81
  Day 365 fold rise | 9.97 (1.093) | 2.00 (5.343)

7. Secondary Outcome: Changes From Baseline in GMFRs Values in SARSCoV- 2 nAbs (Pseudo Neutralization Assay)
Description: as for outcome 4
Time Frame: as for outcome 5
Population: nAb Evaluable Analysis Set - Pseudo Virus
Measure: Geometric Mean (Standard Deviation); unit: Fold rise
Arm/Group | AZD7442: 600mg ONCE / 300mg Q3M | AZD7442: 1200 mg ONCE / 600mg Q6M
Number analyzed (Participants) | 112 | 119
Fold rise
  Day 29 fold rise: number analyzed (Participants) | 88 | 94
  Day 29 fold rise | 18.02 (7.081) | 58.84 (8.473)
  Day 92 fold rise: number analyzed (Participants) | 69 | 85
  Day 92 fold rise | 7.82 (7.270) | 20.38 (8.068)
  Day 121 fold rise: number analyzed (Participants) | 73 | 0
  Day 121 fold rise | 13.13 (8.439) |
  Day 183 fold rise: number analyzed (Participants) | 66 | 80
  Day 183 fold rise | 7.28 (6.954) | 6.90 (7.185)
  Day 212 fold rise: number analyzed (Participants) | 63 | 79
  Day 212 fold rise | 10.28 (6.969) | 14.44 (7.457)
  Day 274 fold rise: number analyzed (Participants) | 59 | 69
  Day 274 fold rise | 7.06 (6.133) | 8.99 (8.271)
  Day 365 fold rise: number analyzed (Participants) | 2 | 67
  Day 365 fold rise | 12.64 (1.251) | 2.84 (8.353)

ADVERSE EVENTS:
Time Frame: Safety data were recorded from the time of the first IMP administration throughout the study for an average safety follow up time of 48.85 weeks. This was shorter than the planned one of 105 weeks due to FDA's request to halt dosing.
Arm/Group | AZD7442: 600mg ONCE / 300mg Q3M | AZD7442: 1200 mg ONCE / 600mg Q6M
All-Cause Mortality (participants affected / at risk) | 0/124 | 1/124
Serious Adverse Events (participants affected / at risk) | 13/124 | 10/124
Other Adverse Events (participants affected / at risk) | 76/124 | 58/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD7442: 600mg ONCE / 300mg Q3M (N=124) | AZD7442: 1200 mg ONCE / 600mg Q6M (N=124)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 2 (2)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (2)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Gastrointestinal anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Focal dyscognitive seizures (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Uraemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD7442: 600mg ONCE / 300mg Q3M (N=124) | AZD7442: 1200 mg ONCE / 600mg Q6M (N=124)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 4 (5)
Nausea (Gastrointestinal disorders) | 4 (8) | 4 (5)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Chills (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 6 (8) | 5 (8)
Injection site pain (General disorders) | 2 (2) | 0 (0)
Injection site pruritus (General disorders) | 1 (1) | 3 (3)
Pain (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Bronchitis (Infections and infestations) | 5 (5) | 0 (0)
Covid-19 (Infections and infestations) | 10 (10) | 12 (13)
Cystitis (Infections and infestations) | 2 (2) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2) | 1 (1)
Herpes zoster (Infections and infestations) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 11 (13) | 7 (7)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Respiratory tract infection viral (Infections and infestations) | 3 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 4 (4)
Urinary tract infection (Infections and infestations) | 7 (7) | 7 (7)
Viral upper respiratory tract infection (Infections and infestations) | 6 (12) | 6 (7)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 3 (3)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Blood pressure increased (Investigations) | 2 (3) | 1 (1)
Blood thrombin increased (Investigations) | 1 (1) | 3 (3)
C-reactive protein increased (Investigations) | 2 (2) | 2 (2)
Troponin increased (Investigations) | 1 (1) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 7 (7) | 1 (1)
Headache (Nervous system disorders) | 8 (8) | 8 (10)
Migraine (Nervous system disorders) | 2 (2) | 1 (1)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 3 (3)
End stage renal disease (Renal and urinary disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 5 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (6)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 5 (5)
Hypotension (Vascular disorders) | 2 (2) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Sponsor terminated the study after review of FDA's request to halt further dosing (30Mar2023) and subjects were terminated prior to 1 year dose given that AZD7442 is not active against >99% of the currently circulating SARS-CoV-2 variants in the USA, the benefit risk assessment may not be favorable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT05375760/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-27): https://cdn.clinicaltrials.gov/large-docs/60/NCT05375760/SAP_001.pdf